CLINICAL TRIAL: NCT03030664
Title: Randomised Controlled Trial With Two Parallel Arms Testing the Effect of L. Reuteri on Bowel Movements in Children Aged 6 Months to 4 Years
Brief Title: Effect of L. Reuteri on Bowel Movements in Children (BIOWELL Study)
Acronym: BIOWELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Camille JUNG, Head of the clinical research department, Centre Hospitalier Intercommunal Creteil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIOWELL; 2016-A00419-42 (Other: ID-RCB)
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Constipation
Keywords: constipation; Lactobacillus reuteri; probiotics
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L.reuteri (Active Comparator): probiotics: L.reuteri produced by Biogaia 5 drops per day: 10exp(8) colony forming unit will be delivered
  Interventions: Dietary Supplement: L.reuteri
- Placebo (Placebo Comparator): Same formulation as probiotics, without active substance. 5 drops per day will be delivered
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: L.reuteri — Each day, at about the same time, the subjects will be given 5 drops (1x10^8 CFU) of the study product in connection with feeding
  Other Names: Lactobacillus reuteri
  Arms: L.reuteri
Drug: Placebo — Same formulation as study product, without probiotics.
  Arms: Placebo

SUMMARY:
A randomized, multicenter, placebo-controlled, double blind study in two parallel groups testing the efficacy of daily oral supplementation with the probiotic L.reuteri DSM17938 compared to placebo in increasing the number of spontaneous bowel movements in infants and children with functional constipation.

DETAILED DESCRIPTION:
Functional constipation in infants up to 4 years of age is defined according to Rome III criteria (Hyman 2006). The diagnose must include 1 month of at least two of the following criteria: two or fewer defecations per week; at least 1 episode per week of incontinence after the acquisition of toilet skills; history of excessive stool retention; history of painful or hard bowel movements; presence of a large faecal mass in the rectum; history of large-diameter stools that may obstruct the toilet.

Accompanying symptoms may include irritability, decreased appetite and/or early satiety. The accompanying symptoms disappear immediately following passage of a large stool.

There is a growing interest for the use of probiotics in functional constipation as research suggests that probiotics could provide beneficial support in the traditional treatment arsenal although the mechanisms of actions are not completely understood.

Wu et al have demonstrated that Lactobacillus reuteri DSM 17938 may have a region-specific intestinal effect on gut motility and therefore could be beneficial in treatment of constipation

Lactobacillus reuteri DSM 17938 has shown significant favourable effects in adults (Ojetti 2014) and young children as described above (Coccorullo 2010, Olgac 2013). These studies require confirmation however. The present clinical study has been designed to strengthen the current available data that L. reuteri DSM 17938 has beneficial effects in infants and young children with functional constipation.

We hypothesize that daily oral supplementation with the probiotic Lactobacillus reuteri DSM 17938 will effectively increase the number of spontaneous bowel movements in infants/children diagnosed with functional constipation according to Rome IV.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 months up to 4 years
* Suffering from functional constipation, as defined by modified Rome III criteria for children aged 4 years or less (Hyman 2006)
* Parent(s) willingness to postpone major changes in the infant feeding mode
* Parent(s) willingness and ability to fill in diary and questionnaires
* Written informed consent from parents
* Stated availability throughout the study period

Exclusion Criteria:

* Chronic illness or major medical problem
* Gastrointestinal disease (including organic cause of constipation and dyschezia or history of severe fecalome)
* Intractable constipation (not responding to conventional treatment for more than 3 months)
* Gastrointestinal surgery (in the year before enrolment)
* Food allergy, lactose or gluten intolerance, as declared by parents
* Use of L. reuteri two weeks before randomisation and throughout the intervention period. If fed with infant formula, it cannot contain L. reuteri.
* Use of antibiotics two weeks before randomisation and throughout the intervention period, both infant/child and lactating mother
* If breastfeeding, use of L reuteri by the mother 2 weeks prior to enrolment
* Conventional treatment for constipation within 2 weeks before enrolment
* Medication that influences gastrointestinal motility
* Mental or behavioral disorders as judged by the investigator

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in number of spontaneous bowel movements | Week 4
  Change in number of spontaneous bowel movements at week 4 compared to baseline evaluated by a bowel habit questionnaire (BQH)

SECONDARY OUTCOMES:
rescue medication | week 4
  Total number of rescue medication during the intervention period
fecal retention | week 4
  number of subjects with 3 or more than 3 stools per week and without fecal retention at the last week of the intervention period
weekly number of spontaneous bowel movements | week 1
  weekly number of spontaneous bowel movements evaluated by the Bowel habit Questionnaire
weekly number of spontaneous bowel movements | week 2
  weekly number of spontaneous bowel movements evaluated by the Bowel habit Questionnaire
weekly number of spontaneous bowel movements | week 3
  weekly number of spontaneous bowel movements evaluated by the Bowel habit Questionnaire
weekly number of spontaneous bowel movements | week 4
  weekly number of spontaneous bowel movements evaluated by the Bowel habit Questionnaire
weekly number of spontaneous bowel movements | week 8
  weekly number of spontaneous bowel movements evaluated by the Bowel habit Questionnaire
Score of QOL | baseline
  Score of quality of life measured using the PedsQL Parent family acute version
Score of QOL | week 4
  Score of quality of life measured using the PedsQL Parent family acute version
Score of QOL | week 8
  Score of quality of life measured using the PedsQL Parent family acute version
Pain during defecation | baseline
  Score of pain during defecation measured using Hick or Wong baker faces
Pain during defecation | week 4
  Score of pain during defecation measured using Hick or Wong baker faces
Pain during defecation | week 8
  Score of pain during defecation measured using Hick or Wong baker faces

CONTACTS AND LOCATIONS:
Overall Officials: Marc BELLAICHE, MD, Principal Investigator — Hopital Universitaire Robert-Debre
Locations (5):
- France (5):
  - CH Sud francilien, Corbeil-Essonnes
  - CHI Creteil, Créteil
  - Hôpital J. Monod - Pavillon Femme Mère Enfant - Le Havre, Le Havre
  - Hôpital Saint Vincent-de-Paul, Lille
  - CHU Robert Debré, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung C, Kalach N, Degas V, Jeridi Y, Bertrand V, Bellaiche M. Effect of L. reuteri on bowel movements in children aged 6 months to 4 years: A double-blind randomized controlled trial. Front Pediatr. 2022 Oct 26;10:997104. doi: 10.3389/fped.2022.997104. eCollection 2022. PMID 36389355